CLINICAL TRIAL: NCT00479128
Title: Phase I Two-Dimensional Dose-Finding Study of Bortezomib in Combination With Gemcitabine/Doxorubicin in Metastatic Surgically Unresectable Urothelial Cancer or Other Solid Tumors
Brief Title: Bortezomib With Gemcitabine/Doxorubicin in Patients With Urothelial Cancer and Other Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0014; NCI-2019-06147 (Registry Identifier: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor; Urethral Cancer
Keywords: Solid Tumor; Bladder Cancer; Ureteral Cancer; Urothelial Cancer; Urethral Cancer; Renal Pelvis Tumor; Bortezomib; Gemcitabine; Doxorubicin; Gemzar; Adriamycin; Velcade; LDP-341; MLN341; PS-341; Gemcitabine Hydrochloride; AD; Hydroxydaunomycin hydrochloride
MeSH Terms: conditions — Urethral Neoplasms; Urinary Bladder Neoplasms; Ureteral Neoplasms | interventions — Bortezomib; Gemcitabine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bortezomib + Gemcitabine + Doxorubicin (Experimental): Starting dose of Bortezomib 0.8 mg/m^2 IV Over 3-5 Seconds. Starting dose of Gemcitabine 225 mg/m^2 IV Up to 90 Minutes. Starting dose of Doxorubicin 12.5 mg/m^2 IV Over 15-30 minutes.
  Interventions: Drug: Bortezomib; Drug: Gemcitabine; Drug: Doxorubicin

INTERVENTIONS:
Drug: Bortezomib — Starting dose: 0.8 mg/m^2 IV Over 3-5 Seconds
  Other Names: Velcade; LDP-341; MLN341; PS-341
Drug: Gemcitabine — Starting dose: 225 mg/m^2 IV Up to 90 Minutes
  Other Names: Gemzar; Gemcitabine Hydrochloride
Drug: Doxorubicin — Starting dose: 12.5 mg/m^2 IV Over 15-30 minutes
  Other Names: Adriamycin; AD; Hydroxydaunomycin hydrochloride

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Gemzar® (gemcitabine) and Adriamycin® (doxorubicin) that can be given together with Velcade® (bortezomib) in patients with urothelial cancer or other solid tumors.

DETAILED DESCRIPTION:
Gemcitabine and doxorubicin are designed to disrupt the growth of cancer cells, which causes cancer cells to start to die. Bortezomib is designed to enter cells and interfere with a substance found inside cells that is responsible for allowing cells to divide. This helps to kill the tumor cells.

If you are found to be eligible to take part in this study, you will receive doses of the study drugs based on when you join the study and how many people have started before you. Two (2) participants will be entered into each dose level. Additional participants may be added at a dose level if it is being well tolerated. The doses will increase until the highest tolerable dose is found.

You will receive the 3 study drugs on the first day of each cycle. You will receive gemcitabine for up to 90 minutes. Next you will receive doxorubicin over 15-30 minutes. Bortezomib will be given last over 3-5 seconds. Every 14 days is considered a study "cycle."

While on study, you will have a complete physical exam before each dose of study drugs. Blood (about 3 teaspoons) will be drawn to check bone marrow and kidney function each week during the first month. The study doctor may decide to draw blood more often, if you are having side effects to the study drugs. Your vital signs will be measured before you receive the study drugs and 1 hour after the infusion.

At the end of Cycle 3, your tumor status will be re-evaluated. You will have CT scans and a bone scan. Blood (about 2 tablespoons) will be drawn for routine tests.

You will be taken off study if the disease gets worse or intolerable side effects occur. If you have stable disease, you may continue receiving therapy as long as your physician feel you are benefiting.

Once you are off-study, you will receive a phone call every 6 months. You will be asked how you are doing, the status of the disease, and if you have had other treatments.

This is an investigational study. Gemcitabine, doxorubicin, and bortezomib are all FDA approved and commercially available. Their use in this study is considered investigational because they have not been approved in patients with urothelial cancer. Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
2. Female patient is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (ie: a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study.
3. All patients must: Have biopsy proven cancer (i.e. solid tumor) for which there is no standard therapy available. If prior history of ischemic heart disease or exposure to > 200 mg/m^2 of doxorubicin, patients must have a measured ejection fraction (either by MUGA, ECHO or ventriculography) of at least 45%. Have preserved hepatic function as shown by AST (SGOT) levels < 2 x the upper limit of normal and an INR (for patients NOT on anticoagulant therapy) of < 1.4. Have normal serum creatinine (<=1.5) or creatinine clearance (measured by Cockcroft -Gault formula) of >= 20 ml/min.
4. All patients must have measurable or evaluable disease. In general, liver and lung lesions should be at least 1 cm, and patients with node-only disease should have lesions of >/= 1.5 cm in greatest dimension. Patients with disease confined to bone may be eligible of a measurable lytic defect is present or a serum marker is elevated (>4 x ULN). The Study Chairman is the final arbiter in questions related to measurability. Patients with a three-dimensional mass or pelvic sidewall fixation on bladder examination under anesthesia are considered to have measurable disease.
5. For the second stage of the Phase I trial, all patients must have histologic demonstration of metastatic or locally unresectable transitional cell carcinoma of the urothelium. Minor components (<50% overall) of variant such as glandular or squamous differentiation, or evolution to more aggressive phenotypes such as sarcomatoid or small cell change are acceptable. However, when these atypical histologies are dominant, other treatment approaches may be more appropriate, and such patients are not eligible.
6. Zubrod performance status </= 2.
7. Patients must have had at least one prior therapy to be eligible for either the first or second stage a) Patients are eligible with any number of prior regimens regardless of what those regimens contained (i.e. prior Bortezomib or combination gemcitabine and adriamycin is acceptable).

Exclusion Criteria:

1. Patient has a platelet count of < 100 x 10^9/L.
2. Patient has an absolute neutrophil count of < 1.2 x 10^9/L.
3. Patient has >/= Grade 2 peripheral neuropathy within 14 days before enrollment.
4. Patient has total bilirubin > 2.5 mg/dL.
5. Patient has hypersensitivity to bortezomib, boron, mannitol, gemcitabine, or doxorubicin. Gemcitabine skin rash that be controlled by short course steroids is allowed.
6. Female subject is pregnant or breast-feeding.
7. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test (Unless there is reasonable certainty that beta-hCG is coming from the tumor). Pregnancy testing is not required for post-menopausal or surgically sterilized women.
8. Patient has received other investigational drugs with 14 days before enrollment.
9. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
10. Patients with significant atherosclerotic disease, as defined by: a) Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or ECG evidence of acute ischemia or active conduction system abnormalities. Any prior ECG abnormality at Screening has to be documented by the investigator as not medically relevant. b) Symptomatic congestive heart failure. c) Claudication limiting activity and d) History of cerebrovascular events within the last year (including TIA).
11. Patient have uncontrolled brain metastases or central nervous system disease.
12. Patients with an active, or likely to become active second malignancy.
13. Patients must be at least 6 weeks out from pelvic irradiation, and must not have more than 10% of bone marrow irradiated.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09-28 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Gemzar + Adriamycin Given with Velcade | Prior to each 2 week cycle

SECONDARY OUTCOMES:
Response of Gemzar + Adriamycin Given with Velcade | 42 days
  Participants be assessed for response on the basis of conventional response criteria for urothelial cancer.
  Tumor status re-evaluated by CT scans and a bone scan.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Siefker-Radtke, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org